CLINICAL TRIAL: NCT06555861
Title: Local Recurrence Prediction of by Texture Analysis Derived From Positron Emission Tomography (PET / CT) Imaging of Non-small Cell Lung Cancer (NSCLC) Treated With Stereotactic Radiotherapy (SBRT)
Brief Title: Local Recurrence Prediction of by Texture Analysis Derived From Positron Emission Tomography (PET / CT) Imaging of Non-small Cell Lung Cancer (NSCLC) Treated With Stereotactic Radiotherapy (SBRT) (Retros MUMOFRAT)
Acronym: MUMOFRAT retro
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC18.0283 - Retros MUMOFRAT
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2018-12

CONDITIONS: Identify FDG PET/CT Parameters Predictive of Local Control
Keywords: PET/CT; Radiomics; Early-stage NSCLC; Stereotactic radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this retrospective multicentric study was to develop and evaluate a prognostic FDG PET/CT radiomics signature in early-stage non-small cell lung cancer (NSCLC) patients treated with stereotactic radiotherapy (SBRT).

ELIGIBILITY:
Inclusion Criteria:

* NSCLC stage I-II treated by SBRT
* PET/CT imaging performed within 60 days of SBRT

Exclusion Criteria:

* Lack of follow-up
* Refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty-seven patients with NSCLC stage I-II and tumours diameters below 5 cm according to the 8th American Joint Committee on Cancer classification, treated with definitive curative SBRT from January 2012 to December 2016 at 4 French institutions (Rennes, Tours, Brest and Nantes) were retrospectively included.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Local Recurrence | Time-to-Event measures up to 5 years
  accuracy

SECONDARY OUTCOMES:
Cancer specific survival | Time-to-Event measures up to 5 years
  accuracy
Distant metastasis free survival | Time-to-Event measures up to 5 years
  accuracy
Recurrence free survival | Time-to-Event measures up to 5 years
  accuracy
Overall survival | Time-to-Event measures up to 5 years
  accuracy

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - ICO, Nantes, Saint Herblain
  - CHRU de Brest, Brest
  - Centre Eugènes Marquis, Rennes
  - CHU de Tours, Tours